CLINICAL TRIAL: NCT03412708
Title: The Effects of Vestibular Rehabilitation Therapy Supported With Virtual Reality on Dizziness and Balance in the Elderly Patients With Dizziness
Brief Title: The Effects of Vestibular Rehabilitation Therapy Supported With Virtual Reality in the Elderly Patients With Dizziness
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Oya Topuz, MD, Professor, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PamukkaleU
Record Dates: First submitted 2018-01-12; First posted 2018-01-26 (Actual); Last update posted 2018-01-26 (Actual); Status verified 2018-01

CONDITIONS: Dizziness; Vestibular Rehabilitation; Virtual Reality
MeSH Terms: conditions — Dizziness

STUDY DESIGN:
Intervention Model Description: Prospective
Who Masked: Outcomes Assessor
Masking Description: Single blind
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vestibular Rehabilitation (Active Comparator): Vestibular Rehabilitation Program Exercises for Eye Movements: Smooth- Pursuit Eye Movements and Saccadic eye movements Exercises for Gaze Stability : Training of Vestibulo-ocular reflex and Cervico-ocular reflex Exercises for Postural Stability: In sitting or standing up position and walking
  Duration of treatment: 3 weeks. Number of sessions: 15 Session frequency: 5 times a week. Session duration: 2 sets of 15 minutes, with a 5 minute break between sets, for a total of 35 minutes.
  Interventions: Other: Vestibular Rehabilitation supported with Virtual Reality
- Vestibular Rehabilitation supported with Virtual Reality (Experimental): Patients will perform the exercises in a virtual reality environment using a virtual reality goggle and a smartphone.The virtual environments consist of 2 media provided by the videos taken with a 360 camera . 1) A square with people moving, noise and traffic and 2) A supermarket where the shelves are full. Exercises conducted while sitting and standing on a soft ground will happen in the 1st environment, and the ones on the treadmill will happen in the 2nd environment.
  Exercises for Eye Movements: Smooth- Pursuit Eye Movements and Saccadic eye movements Exercises for Gaze Stability : Training of Vestibulo-ocular reflex and Cervico-ocular reflex Exercises for Postural Stability: In sitting or standing up position and walking
  Duration of treatment: 3 weeks. Number of sessions: 15 Session frequency: 5 times a week. Session duration: 2 sets of 15 minutes, with a 5 minute break between sets, for a total of 35 minutes.
  Interventions: Other: Vestibular Rehabilitation supported with Virtual Reality

INTERVENTIONS:
Other: Vestibular Rehabilitation supported with Virtual Reality — Patients will perform the supervised vestibular exercises in virtual reality environment using a virtual reality goggle (Samsung Gear VR SM323) and a smartphone (Samsung Galaxy S7). The virtual environments consist of 2 media provided by the videos taken with a 360 camera (Samsung Gear 360). 1) A square with people moving, noise and traffic and 2) A supermarket where the shelves are full.

SUMMARY:
Objective: To investigate the effect of vestibular rehabilitation exercises supported with virtual reality using virtual glasses technology on dizziness, static and dynamic balance, functional mobility, fear of falling, anxiety and depression in the short term (3 weeks) in the elderly with dizziness.

DETAILED DESCRIPTION:
INTRODUCTION:

Dizziness, is a condition that includes spatial orientation and motion perception disorder symptoms such as swivel illusion or sensation of instability, which can affect gaze stability, posture and walking. This problem is seen in about 30% of the elderly living in society and the prevalence increases with age (1). Patients with history of dizziness have limitations in daily activities, increased fear of falling, increased anxiety and depression, decreased quality of life, and increased risk of falls (2,3).

It has been shown that vestibular rehabilitation programs including postural control and balance exercises as well as recurrent head, eye, and trunk movements have positive effects on dizziness, balance and falling risk in the elderly (4,5).

Exercise programs are often performed in the clinical setting or at home, and participation in the exercise program of real-life environments such as a street, supermarket, park, workplace, where traffic is available can make a difference in patient motivation and exercise effectiveness. Positive effects on walking, postural control, balance and mobility in the elderly have been reported with exercises in the form of interactive games such as "Nintendo Wii", "Balance Rehabilitation Unit", dance video games where virtual reality technologies are used (6-10). There was no study investigating the effects of virtual reality created by virtual glasses and smartphone technology, on balance, functional mobility, falling risk, anxiety and depression in the elderly.

The objective of this study is to investigate the effect of vestibular rehabilitation exercises supported with virtual reality using virtual glasses technology on dizziness, static and dynamic balance, functional mobility, fear of falling, anxiety and depression in the short term (3 weeks) in the elderly with dizziness.

METHOD:

Research Design:

Single-blind, randomized, controlled, single-center, prospective, experimental study in patients aged 65 years and older who applied to the otorhinolaryngology clinic with dizziness complaint and 6-month follow-up period.

Target Research Group: Patients 65 years of age or older who meet the inclusion criteria below.

Inclusion Criteria: 1) Living in society 2) Being able to stand up and walk by themselves, without needing a supporting device 3) Applying to the otorhinolaryngology clinic with dizziness complaint. Patients with any of the exclusion criteria listed below will be excluded from the study.

Exclusion Criteria: 1) Presence of cognitive dysfunction 2) Presence of musculoskeletal or systemic disease that prevents exercise. 3) Having an exercise program in the last 6 months, 4) Presence of psychiatric or neurological diseases that affect cooperation and cognitive functions in their history, 5) Presence of neurological disease that affects balance in their history, 6) Positive Dix-Hallpike test, 7) Patients with a Vit D level lower than 30 ng /ml.

Beginning Screening Assessments are ,illness inquiry, inquiring about used medication, cigarette and alcohol, history of falling.

The following questions were asked about the fall of the patient and their answers were recorded.

How many times did you fall in the last 6 months? Where did you fall? How did you fall? Were you injured? Were you admitted to the hospital?

Assessment of Cognitive Function by Mini Mental Test:

It was first published by Folstein and his friends. The test is a short, useful and standardized tool that can be used when assessing the cognitive level globally. The orientation is made up of eleven items grouped under five main headings as recording memory, attention and calculation, recall and language, and is evaluated over the total score of 30 (11). In this study, revised Mini Mental State Scale, whose Turkish validity and reliability studies were done by Keskinoğlu et al., was used in educated and uneducated elderly. Cut-off value was accepted as 24 for educated and 19 for uneducated elderly, as indicated by the researchers (12).

Assessing eye movements and visual acuity:

Eye movements: They were asked to make eye movements in all directions.

Smooth pursuit eye movements:

The patient was asked to watch the index finger of the examiner slowly moving up or down, left or right, with their eye. The patient must be able to see the index finger clearly, the finger should not move more than 60 degrees from one side to the other, and the speed should not be more than 40 degrees per second.

Saccadic eye movements:

The patient was asked to look at the fingers separated from each other by vertical and horizontal planes at a distance of 30 cm. During this time, attention was paid to latency, speed, accuracy and parallelism (conjugation) in the movement of the eyes.

Visual Acuity:

Assessed using a Snellen Chart.

Somatosensorial assessment:

Lower extremity muscle strength Lower extremity muscle strength was assessed with Chair Stand Test. This test was performed by Jones et al. and has been shown to be a valid and reliable measure of the proximal muscle strength of the lower extremities in elderly individuals. In the starting position the person is sitting on a chair without armrests and with their back upright, their arms crossed in front of their chest and their feet on the floor. With the start command, the person does a full standing position and is seated again, the total number of full stands in 30 seconds constitutes their score (13).

Lower extremity sense:

On the lower extremity sensory examination, the light touch sensation was assessed by cotton, the pain sensation by a needle, and the deep sensation by the sensation of the thumb position.

Cerebellar Assessment:

Finger - Nose Test The patient touches their nose with their index finger after touching the index finger of the doctor sitting opposite them. While repeating this movement in succession, the physician changes the position of his finger every time. The results were scored as successful / unsuccessful.

Knee - Heel Test It is examined with the patient laying on their back. After the patient touches their knee with their heel, they lower the foot down on a straight line along the tibia bone. After repeating this movement several times, they do the same with the other foot. The results were scored as successful / unsuccessful.

Alternating Movement Tests The patient is made to do quick alternating movements. The patient opens a hand with the palm up. The back of the other hand and the palmar face touch the open palm with rapid repetitive pronation-supination movements. The results were scored as successful / unsuccessful.

Pulse:

Blood pressure:

Orthostatic hypotension:

Postural blood pressure measurement; the first blood pressure was measured after they had been laying on their back for at least five minutes, the second blood pressure was measured as soon as they stood up and third blood pressure was measured after standing on their feet and waiting for three minutes with a manometer. A fall of 20mmHg relative to the lying position in the systolic blood pressure after standing on their feet and after standing for three minutes was considered significant for orthostatic hypotension (14).

Vit D Level:

Calculation of Sample Size:

The sample size was calculated as the minimum number of subjects required for each of the arms so that a difference of 3.73 units between the two group averages in the Berg Balance Scale (Type 1 error: 0,05, Type 2 error: 0,20) could be significant according to the results of the previous study. The number of subjects in each group will be a minimum of 16(15).

Randomisation and treatment:

Patients who meet the inclusion criteria after initial screening and do not have exclusion criteria will be divided into two groups by layered block randomization and 2 different treatment protocols will be applied. Patients were planned to be included so that at least 16 patients would be in each group.

Group 1: Supervised vestibular rehabilitation program in clinical setting. Group 2: Supervised vestibular rehabilitation program supported with virtual reality

For both groups; Duration of treatment: 3 weeks. Number of sessions: 15 Session frequency: 5 times a week. Session duration: 2 sets of 15 minutes, with a 5 minute break between sets, for a total of 35 minutes.

Patients who do not attend at least 3 sessions in the same week will be dropped from the study.

Patients in Group 2 will perform the exercises in a virtual reality environment using a virtual reality goggle (Samsung Gear VR SM323) and a smartphone (Samsung Galaxy S7). The virtual environments consist of 2 media provided by the videos taken with a 360 camera (Samsung Gear 360). 1) A square with people moving, noise and traffic and 2) A supermarket where the shelves are full. Exercises conducted while sitting and standing on a soft ground will happen in the 1st environment, and the ones on the treadmill will happen in the 2nd environment.

During the exercises, assisted ambulation system (Biodex Free Step SAS) will be used to ensure the safety of the patient and to prevent falls.

All patients will be trained initially by a physician for 30 minutes, including a definition of fall, definition of prevention, risk factors, information on prevention, and recommendations for preventing falls.

Vestibular Rehabilitation Program

2 sets of 15 minutes; each set will include the following exercises for a total of a 35 minute program.

Exercises for Eye Movements

Smooth- Pursuit Eye Movements:

The patient is asked to move their eyes at first slowly and then quickly in horizontal and vertical directions (10 times). In the 1st week while sitting, in the 2nd week while standing and in the 3rd week while standing on a soft ground.

Saccadic eye movements:

The patient is asked to focus by moving their eyes 1 time per second to 2 targets 30 cm away from each other (10 times). Motion is applied in horizontal and vertical directions. While sitting on the 1st week, standing on the 2nd week, and standing on soft ground for the 3rd week.

Exercises for Gaze Stability

Training of Vestibulo-ocular reflex:

1. The patient is asked to move their head first in horizontal, then in vertical directions for 1 minute, focusing on a fixed object. While sitting on the 1st week, standing on the 2nd week, and standing on soft ground for the 3rd week.
2. The patient is asked to move their head first in horizontal, then in vertical directions for 1 minute, focusing on a moving object. While sitting on the 1st week, standing on the 2nd week, and standing on soft ground for the 3rd week.

Training of Cervico-ocular reflex The patient sitting on a rotating chair is asked to move their torso to the right and left, keeping his head steady by focusing on a fixed object (10 times). It is conducted in the 1st and 2nd weeks.

Exercises for Postural Stability

Standing up:

1. Week:

   Bend forward and side to side while sitting, pass from sitting position to standing position and back to sitting position (10 times), standing in various positions (feet together, tandem position) (15 sec), marching in place (10 times) is requested.
2. Week:

   Bending their body front and back, and to their sides (10 front and back, 10 to the sides) while standing, standing in various positions (feet together, tandem position) (15 sec), marching in place (10 times) is requested.
3. Week The exercises in the 2nd week is conducted on soft ground.

Walking:

Patients conduct their exercises while walking at a pace of 1.6km/h on the treadmill.

1. Week:

   They are asked to walk forward on the treadmill (1 min)
2. Week:

   They are asked to walk on the treadmill while moving their head left-right, front-back (1 min)
3. Week:

They are asked to walk on the treadmill while focusing on a fixed object and moving their heads first horizontally and then vertically (1 min)

Assessment Parameters

Dizziness Assessment

Vertigo Symptom Scale (Short form):

It is a questionnaire consisting of 15 items evaluating the frequency of dizziness and / or unbalance and accompanying autonomic and anxiety symptoms within the last 1 month. Each item is scored between 0-4 and the scores of all items are summed to obtain the symptom severity score. The total score is between 0 and 60, higher scores indicate a more serious problem. A total score of 12 or more indicates severe dizziness. The scale consists of 8 items related to vertigo-balance, scored between 0-32 points (VSS-V), and 7 items related to autonomic-anxiety symptoms and 2 scales scored between 0-28 points (VSS-A) (16,17). The validity and reliability studies of the Turkish version were made by Yanık et al. (18).

Dizziness Disability Inventory:

The Dizziness Disability Inventory (DDI), developed to measure disability in patients with dizziness and available for follow-up, is a questionnaire consisting of 25 questions about the physical, functional, and emotional state of the patient. There are nine items each that determine the emotional state and functional status and seven items that determine the physical function. If the answers to the questions are "yes", they are scored as four points, "sometimes" as two points, and "no" as zero points. The maximum score for the emotional and functional subgroups is 36, and for the physical function subgroup the maximum score is 28, with a maximum score of 100 in total. The minimum score for all subgroups and total score is zero. High score indicates more disability (19). The validity and reliability studies of the Turkish version were made by Ellialtıoğlu and their colleagues (20).

Balance Assessment

Berg Balance Test:

The Berg balance test (BBT), which was developed by Berg et al. in 1989 and proved to be valid and reliable in 1992, was used as a clinical balance test. This test includes activities such as unsupported seating, standing from a seating position, standing without support, picking up an item from the floor, turning 360 degrees, looking back over the shoulder, and transferring from the bed to the chair. In BBT, the level of qualification for each item is scored from zero to four, where 0 means "can not do it"; and 4 means "can do it independently and safely". The total maximum score is 56 and the higher scores show a better balance (21). Şahin et al. showed that the Turkish version of the Berg balance test was a reliable and valid scale for assessing balance in elderly adults (22).

Dynamic Posturography Biodex Balance System (Biodex, Inc., Shirley, New York) was used to evaluate the dynamic balance in elderly subjects (23,24). Postural stability tests and the risk of falls (General Stability Index, Medio-lateral Stability Index, Antero-posterior Stability Index, Falling Risks Index) were calculated. There is a balance platform of this system in relation to a computer software that allows moving, balanced, objective evaluation of the system, which can be tilted up to 20 ° at a 360 ° range of motion. The overall stability score refers to the balance ability of the person in general and high values indicate that the balance is bad. Patients are tested on the platform at the 8th level, with the eyes open and on both feet, while the feet are naked and the person is in the most comfortable position where they can keep their balance, their knees are at the slightest flexion (15º). After a 20-second trial test, each person was subjected to three 20-second tests. A 10-second rest period was provided between each test, and as a result, averages of these three tests were obtained.

Functional Mobility Assessment

TUG:

Timed Up&Go (TUG) test was used to assess functional mobility. In this test the elapsed time is measured in seconds for the individual to get up from the sitting position, walk a three meter distance and return. During the test, the standard chair with armrests should have a tape, cone or other clear marker indicating the end of the distance and the person should be wearing walking shoes they are used to and if they use a supportive device such as a walker or crutches, this should be noted and also used during the test (25).

Assessment of fear of falling:

International Falls Efficacy Scale:

The test described by Yardley et al. in 2005 consists of 16 questions that assess patients' anxiety about the possibility of falls during their daily activities. Each question is scored between 0-4 in itself (26). The validity and reliability study in Turkish for the elderly population was conducted (27).

Anxiety/Depression Assessment Geriatric Depression Scale To assess depression, we used Geriatric Depression Scale (GDS) developed by Yesavage and colleagues to screen for depression in the elderly population. The scale consists of a total of thirty closed-ended questions. The answers are calculated as "1" point for each question if answered in a depressed way, and the sum of these points and the total score are calculated. The high scores indicate depressive characteristics. The total score is thirty, with the scores meaning no depression between 0-11, possible depression between 11-14, and definite depression for 14 and over (28). The validity and reliability of the GDS has been proven by translating it into Turkish by Ertan and his colleagues (29).

Hamilton Anxiety Assessment Scale:

This scale, developed by Hamilton, questions the anxiety severity, psychological and somatic symptoms. In the 14 questions, topics such as anxious temperament, tension, fear, insomnia, intellectual status, depressive temperament, body symptoms, somatic symptoms, cardiovascular symptoms, respiratory symptoms, gastrointestinal symptoms, genitourinary symptoms, autonomic symptoms and behaviours during the interview are questioned. When each of the 14 items are assessed, a score of 0-4 is given (0=none, 1=mild, 2=medium, 3=severe, 4=very severe) and the patients are evaluated based on the scores they receive in the overall total. The higher the score, the higher the severity of anxiety. The total score is between 0-56, below 17 is mild, between 18-24 is moderate and 25-30 is severe (30). Reliability and validity studies in Turkey were made by Yazıcı and his colleagues (31).

ELIGIBILITY:
Inclusion Criteria:

1. Living in society
2. Being able to stand up and walk by themselves, without needing a supporting device
3. Consulting an otolaryngologist with the complaint of dizziness.

Exclusion Criteria:

1. Presence of cognitive dysfunction
2. Presence of musculoskeletal or systemic disease that prevents exercise.
3. Having an exercise program in the last 6 months,
4. Presence of psychiatric or neurological diseases that affect cooperation and cognitive functions in their history,
5. Presence of neurological disease that affects balance in their history,
6. Positive Dix-Hallpike test,
7. Patients with a Vit D level lower than 30 ng /ml.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2017-05-23 (Actual); Primary Completion 2018-11 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Vertigo Symptom Scale (Short form) | 3 weeks
  Vertigo Symptom Scale (Short form) is a questionnaire consisting of 15 items evaluating the frequency of dizziness and / or unbalance and accompanying autonomic and anxiety symptoms within the last 1 month.
Dizziness Handicap Inventory | 3 weeks
  The Dizziness Handicap Inventory , developed to measure disability in patients with dizziness and available for follow-up, is a questionnaire consisting of 25 questions about the physical, functional, and emotional state of the patient.
Berg Balance Test | 3 weeks
  Berg Balance Test includes activities such as unsupported seating, standing from a seating position, standing without support, picking up an item from the floor, turning 360 degrees, looking back over the shoulder, and transferring from the bed to the chair.
Dynamic Posturography | 3 weeks
  Biodex Balance System (Biodex, Inc., Shirley, New York) was used to evaluate the dynamic balance in elderly subjects Postural stability tests and the risk of falls (General Stability Index, Medio-lateral Stability Index, Antero-posterior Stability Index, Falling Risks Index) were calculated.

SECONDARY OUTCOMES:
Timed Up&Go (TUG) test | 3 weeks
  Timed Up&Go (TUG) test was used to assess functional mobility.
International Falls Efficacy Scale | 3 weeks
  International Falls Efficacy Scale: The test consists of 16 questions that assess patients' anxiety about the possibility of falls during their daily activities.
Geriatric Depression Scale | 3 weeks
  Geriatric Depression Scale consists of a total of thirty closed-ended questions. The answers are calculated as "1" point for each question if answered in a depressed way, and the sum of these points and the total score are calculated.
Hamilton Anxiety Assessment Scale | 3 weeks
  Hamilton Anxiety Assessment Scale questions the anxiety severity, psychological and somatic symptoms. severity of anxiety

CONTACTS AND LOCATIONS:
Locations (1):
- Pamukkale University Faculty of Medicine, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Fernandez L, Breinbauer HA, Delano PH. Vertigo and Dizziness in the Elderly. Front Neurol. 2015 Jun 26;6:144. doi: 10.3389/fneur.2015.00144. eCollection 2015. PMID 26167157
- [Background] Salles N, Kressig RW, Michel JP. Management of chronic dizziness in elderly people. Z Gerontol Geriatr. 2003 Feb;36(1):10-5. doi: 10.1007/s00391-003-0141-x. PMID 12616402
- [Background] Lo AX, Harada CN. Geriatric dizziness: evolving diagnostic and therapeutic approaches for the emergency department. Clin Geriatr Med. 2013 Feb;29(1):181-204. doi: 10.1016/j.cger.2012.10.004. PMID 23177607
- [Background] Yang XJ, Hill K, Moore K, Williams S, Dowson L, Borschmann K, Simpson JA, Dharmage SC. Effectiveness of a targeted exercise intervention in reversing older people's mild balance dysfunction: a randomized controlled trial. Phys Ther. 2012 Jan;92(1):24-37. doi: 10.2522/ptj.20100289. Epub 2011 Oct 6. PMID 21979272
- [Background] Jung JY, Kim JS, Chung PS, Woo SH, Rhee CK. Effect of vestibular rehabilitation on dizziness in the elderly. Am J Otolaryngol. 2009 Sep-Oct;30(5):295-9. doi: 10.1016/j.amjoto.2008.06.013. Epub 2009 Feb 6. PMID 19720245
- [Background] Duque G, Boersma D, Loza-Diaz G, Hassan S, Suarez H, Geisinger D, Suriyaarachchi P, Sharma A, Demontiero O. Effects of balance training using a virtual-reality system in older fallers. Clin Interv Aging. 2013;8:257-63. doi: 10.2147/CIA.S41453. Epub 2013 Feb 28. PMID 23467506
- [Background] Toulotte C, Toursel C, Olivier N. Wii Fit(R) training vs. Adapted Physical Activities: which one is the most appropriate to improve the balance of independent senior subjects? A randomized controlled study. Clin Rehabil. 2012 Sep;26(9):827-35. doi: 10.1177/0269215511434996. Epub 2012 Feb 9. PMID 22324055
- [Background] Pichierri G, Murer K, de Bruin ED. A cognitive-motor intervention using a dance video game to enhance foot placement accuracy and gait under dual task conditions in older adults: a randomized controlled trial. BMC Geriatr. 2012 Dec 14;12:74. doi: 10.1186/1471-2318-12-74. PMID 23241332
- [Background] Laver K, George S, Ratcliffe J, Quinn S, Whitehead C, Davies O, Crotty M. Use of an interactive video gaming program compared with conventional physiotherapy for hospitalised older adults: a feasibility trial. Disabil Rehabil. 2012;34(21):1802-8. doi: 10.3109/09638288.2012.662570. Epub 2012 Mar 12. PMID 22409245
- [Background] Szturm T, Betker AL, Moussavi Z, Desai A, Goodman V. Effects of an interactive computer game exercise regimen on balance impairment in frail community-dwelling older adults: a randomized controlled trial. Phys Ther. 2011 Oct;91(10):1449-62. doi: 10.2522/ptj.20090205. Epub 2011 Jul 28. PMID 21799138
- [Background] Folstein MF, Folstein SE, McHugh PR. "Mini-mental state". A practical method for grading the cognitive state of patients for the clinician. J Psychiatr Res. 1975 Nov;12(3):189-98. doi: 10.1016/0022-3956(75)90026-6. No abstract available. PMID 1202204
- [Background] Keskinoglu P, Ucku R, Yener G, Yaka E, Kurt P, Tunca Z. Reliability and validity of revised Turkish version of Mini Mental State Examination (rMMSE-T) in community-dwelling educated and uneducated elderly. Int J Geriatr Psychiatry. 2009 Nov;24(11):1242-50. doi: 10.1002/gps.2252. PMID 19337986
- [Background] Jones CJ, Rikli RE, Beam WC. A 30-s chair-stand test as a measure of lower body strength in community-residing older adults. Res Q Exerc Sport. 1999 Jun;70(2):113-9. doi: 10.1080/02701367.1999.10608028. PMID 10380242
- [Background] Kaufmann H. Consensus statement on the definition of orthostatic hypotension, pure autonomic failure and multiple system atrophy. Clin Auton Res. 1996 Apr;6(2):125-6. doi: 10.1007/BF02291236. No abstract available. PMID 8726100
- [Background] Karahan AY, Tok F, Taskin H, Kucuksarac S, Basaran A, Yildirim P. Effects of Exergames on Balance, Functional Mobility, and Quality of Life of Geriatrics Versus Home Exercise Programme: Randomized Controlled Study. Cent Eur J Public Health. 2015 Nov;23 Suppl:S14-8. doi: 10.21101/cejph.a4081. PMID 26849537
- [Background] Yardley L, Masson E, Verschuur C, Haacke N, Luxon L. Symptoms, anxiety and handicap in dizzy patients: development of the vertigo symptom scale. J Psychosom Res. 1992 Dec;36(8):731-41. doi: 10.1016/0022-3999(92)90131-k. PMID 1432863
- [Background] Yardley L, Beech S, Zander L, Evans T, Weinman J. A randomized controlled trial of exercise therapy for dizziness and vertigo in primary care. Br J Gen Pract. 1998 Apr;48(429):1136-40. PMID 9667087
- [Background] Yanik B, Kulcu DG, Kurtais Y, Boynukalin S, Kurtarah H, Gokmen D. The reliability and validity of the Vertigo Symptom Scale and the Vertigo Dizziness Imbalance Questionnaires in a Turkish patient population with benign paroxysmal positional vertigo. J Vestib Res. 2008;18(2-3):159-70. PMID 19126986
- [Background] Jacobson GP, Newman CW. The development of the Dizziness Handicap Inventory. Arch Otolaryngol Head Neck Surg. 1990 Apr;116(4):424-7. doi: 10.1001/archotol.1990.01870040046011. PMID 2317323
- [Background] Ellialtıoğlu A, Karan A, İşsever H, Aksoy C. Validity and reliability of Turkish version of Dizziness Handicap Inventory (DHI). XVIII National Physical Medicine and Rehabilitation Congress, May 12-17, 2001, Antalya, Program and Abstract Book; 2001. p. 131
- [Background] Berg KO, Maki BE, Williams JI, Holliday PJ, Wood-Dauphinee SL. Clinical and laboratory measures of postural balance in an elderly population. Arch Phys Med Rehabil. 1992 Nov;73(11):1073-80. PMID 1444775
- [Background] Sahin F, Yilmaz F, Ozmaden A, Kotevolu N, Sahin T, Kuran B. Reliability and validity of the Turkish version of the Berg Balance Scale. J Geriatr Phys Ther. 2008;31(1):32-7. doi: 10.1519/00139143-200831010-00006. PMID 18489806
- [Background] Baldwin, S.L., T.W. VanArnam,L.L. Ploutz-Snyder. Reliability of dynamic bilateral postural stability on the Biodex Stability System in older adults. Medicine & Science in Sports & Exercise, 2004(36):30
- [Background] Parraca, J.A., Olivares, P.R., Carbonell-Baeza, A., Aparicio, V.A., Adsuar, J.C., Gusi, N. Test-retest reliability of Biodex Balance SD on physically active old people. J Hum Sport Exerc. 2011;6:444-451
- [Background] Podsiadlo D, Richardson S. The timed "Up & Go": a test of basic functional mobility for frail elderly persons. J Am Geriatr Soc. 1991 Feb;39(2):142-8. doi: 10.1111/j.1532-5415.1991.tb01616.x. PMID 1991946
- [Background] Yardley L, Beyer N, Hauer K, Kempen G, Piot-Ziegler C, Todd C. Development and initial validation of the Falls Efficacy Scale-International (FES-I). Age Ageing. 2005 Nov;34(6):614-9. doi: 10.1093/ageing/afi196. PMID 16267188
- [Background] Ulus Y, Durmus D, Akyol Y, Terzi Y, Bilgici A, Kuru O. Reliability and validity of the Turkish version of the Falls Efficacy Scale International (FES-I) in community-dwelling older persons. Arch Gerontol Geriatr. 2012 May-Jun;54(3):429-33. doi: 10.1016/j.archger.2011.06.010. Epub 2011 Aug 9. PMID 21831462
- [Background] Yesavage JA, Brink TL, Rose TL, Lum O, Huang V, Adey M, Leirer VO. Development and validation of a geriatric depression screening scale: a preliminary report. J Psychiatr Res. 1982-1983;17(1):37-49. doi: 10.1016/0022-3956(82)90033-4. PMID 7183759
- [Background] Ertan T, Eker E, Sar V. Geriatrik Depresyon Ölçegi'nin Türk Yaslı Nüfusunda Geçerlilik ve Güvenilirligi. Nöropsikiyatri Arsivi 1997; 34(2): 62-71
- [Background] HAMILTON M. The assessment of anxiety states by rating. Br J Med Psychol. 1959;32(1):50-5. doi: 10.1111/j.2044-8341.1959.tb00467.x. No abstract available. PMID 13638508
- [Background] Yazıcı MK, Demir B, Tanrıverdi N, Karaağaoğlu E, Yolaç¸ P. Hamilton Anksiyete Değerlendirme Ölçeği Değerlendiriciler Arası Güvenilirlik ve Geçerlilik Çalışması. Türk Psikiyatri Dergisi 1998;9:114-7